CLINICAL TRIAL: NCT04611243
Title: Lung Function, Exercise Capacity, and Serology Responses in Patients With COVID-19
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The University of Hong Kong (Other); Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Prof David Shu Cheong Hui, Professor, Chinese University of Hong Kong
Other Study IDs: 2020.229
Record Dates: First submitted 2020-06-29; First posted 2020-11-02 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Lung Function; Exercise Capacity; Quality of Life; Covid19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine; Vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be taken for serology testing and T cell response after discharge, 6, 12, 18 and 24 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- COVID survivors
- Vaccination with CoronaVac vaccine
  Interventions: Biological: Vaccination with Coronavac vaccine
- Vaccination with BionTech vaccine
  Interventions: Biological: Vaccination with BionTech Vaccine
- third dose vaccination with CoronaVac vaccine: We propose to invite 80 participants who have already completed the 2 doses vaccination of CoronaVac with low level of neutralizing antibody at 1-month post-vaccination to join this additional study. They will be randomized to receive a booster dose of Coronavac or BionTech in equal numbers (n=40 each group).
  Interventions: Biological: third dose vaccination with CoronaVac vaccine
- third dose vaccination with BionTech vaccine: We propose to invite 80 participants who have already completed the 2 doses vaccination of CoronaVac with low level of neutralizing antibody at 1-month post-vaccination to join this additional study. They will be randomized to receive a booster dose of Coronavac or BionTech in equal numbers (n=40 each group).
  Interventions: Biological: third dose vaccination with BionTech vaccine

INTERVENTIONS:
Biological: third dose vaccination with CoronaVac vaccine — Healthy individuals with low antibody levels after 2 doses of CoronaVac vaccine to receive one additional dose of CoronaVac vaccine
  Groups: third dose vaccination with CoronaVac vaccine
Biological: third dose vaccination with BionTech vaccine — Healthy individuals with low antibody levels after 2 doses of CoronaVac vaccine to receive one additional dose of BionTech vaccine
  Groups: third dose vaccination with BionTech vaccine
Biological: Vaccination with Coronavac vaccine — Healthy individuals to receive Coronavac vaccine 2 doses, 21 days apart
  Groups: Vaccination with CoronaVac vaccine
Biological: Vaccination with BionTech Vaccine — Healthy individuals to receive BionTech vaccine 2 doses, 21 days apart
  Groups: Vaccination with BionTech vaccine

SUMMARY:
(a) Objectives

1. To assess the full lung function, exercise capacity, quality of life in patients with COVID-19 over 2 years.
2. To assess the longevity of the serology response to SARS-CoV2.
3. To investigate the association of the neutralization titer in plasma from different vaccinated cohorts to its protection of infection using in vivo model
4. To investigate the SARS-CoV-2 specific cellular and humoral immunities as well as their determinant factors from community subjects who have received different types of COVID-19 vaccines.
5. To assess the third booster dose for subjects who have poor antibody response despite having received two doses of CoronaVac (Sinovac)

DETAILED DESCRIPTION:
The health conditions of adults (N=300) who recovered from varying severity of COVID-19 will be assessed and their blood are collected at 6, 12, 24 and 36 months after discharge. The assessment package includes: lung function tests, 6-min walk distance, chest radiographs/CT, and SF36 General Health questionnaire. Blood samples from community cohorts will be collected from before and up to 36 months after receiving one of the three COVID-19 vaccines (N=200 per vaccine type). The kinetics of SARS-CoV-2 specific humoral and cellular immunities from both convalescent and vaccinated cohorts are determined by neutralization assay and by measuring specific T cell responses upon stimulation of SARS-CoV-2 specific peptide library respectively. The antiviral level of the human plasma with various neutralization titer collected from different vaccinated cohorts will be tested in mouse model and ADCC assay.

ELIGIBILITY:
Inclusion Criteria: Patients who have been discharged from hospital following treatment for COVID-19 -

Exclusion Criteria: Unwilling to be follow up

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (about 80) who have been discharged following treatment for COVID-19 will be followed up at the Prince of Wales Hospital at 4 weeks after discharge, 6, 12, 18 and 24 months.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-05-22 (Actual); Primary Completion 2025-08-18 (Estimated); Study Completion 2026-02-17 (Estimated)

PRIMARY OUTCOMES:
spirometry | 3 years
  FEV1 and FVC
Lung volume | 3 years
  Litres
6 minute walk distance | 3 years
  meters

SECONDARY OUTCOMES:
quality of life by SF36 questionnaire | 3 years
  scores in all domains
serology and T cell response | 3 years
  titers

CONTACTS AND LOCATIONS:
Overall Officials: David S Hui, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
data pending

REFERENCES:
- [Derived] Chan KKP, Ng SSS, Lui GCY, Leung HS, Wong KT, Chu WCW, Chan TO, Yiu KYS, Tso EYK, To KW, Ngai JCL, Yip TWH, Lo RLP, Ng JKC, Ko FWS, Hui DSC. Comparison of the 12-month impact of COVID-19 and SARS on physiological capacity and health-related quality of life. BMC Pulm Med. 2023 Nov 14;23(1):441. doi: 10.1186/s12890-023-02750-8. PMID 37964259